CLINICAL TRIAL: NCT00400296
Title: A Multiple Ascending Dose (MAD) Study of R547 Administered as an Intravenous Infusion on a Weekly Schedule in Patients With Advanced Solid Tumors
Brief Title: A Study of R547 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP18378
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG547

INTERVENTIONS:
Drug: RG547 — Administered iv on days 1 and 8 of a 3 week cycle at escalating doses to successive groups of patients until MTD is reached.

SUMMARY:
This single arm study will determine the maximum tolerated dose, and recommended dose for further development, of R547, in patients with advanced solid tumors. Groups of patients will receive ascending doses of R547 as weekly intravenous infusions administered over a) 90 minutes and b) 180 minutes, on days 1 and 8 of a 21 day cycle. In the absence of dose-limiting toxicity following the starting dose, incremental dose-escalations will be allowed in subsequent cohorts of patients until the maximum tolerated dose is reached. The anticipated time on study treatment is until disease progression or dose-limiting toxicity, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* locally advanced or metastatic solid tumors;
* measurable or evaluable disease.

Exclusion Criteria:

* prior chemotherapy, radiotherapy or immunotherapy within 3 weeks of start of study;
* prior history of CNS metastases with disease progression;
* patients taking strong inhibitors and/or inducers of CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters. | Throughout study

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic profiles of R547 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Aurora, Colorado
  - New Brunswick, New Jersey
  - Charlotte, North Carolina
  - Houston, Texas

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148